CLINICAL TRIAL: NCT05417698
Title: Evaluation of Lifestyle Modification on Cardiovascular Risk in Overweight and Obese Postmenopausal Women: a Ghrelin-mediated Response
Brief Title: Evaluation of Lifestyle Modification on Cardiovascular Risk
Acronym: GHRexD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIO 035-20
Record Dates: First submitted 2022-04-11; First posted 2022-06-14 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Menopause; Cardiovascular Diseases; Obesity; Type2diabetes
Keywords: Ghrelin; Postmenopause
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Obesity | interventions — Exercise; Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Randomised-controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise only (Ex only) (Experimental): Participants in the "Exercise only" group will be performing home-based, equipment-free HIIT exercise for 20 minutes, 3 times a week for the duration of the 8-weeks, achieving ≥80% of predicted heart rate maximum (HRmax; 220-age) during the high-intensity intervals. Participants are also required to exercise at least 17 out of 20 on the Rate of Perceived Exertion (RPE) scale.
  Interventions: Other: Exercise Only (Ex only)
- Exercise and Mediterranean Diet (Ex + MedDiet) (Experimental): Participants in Ex+MedDiet arm will be required to adhere to a non-caloric restrictive Mediterranean diet throughout the 8-weeks according to a Mediterranean diet booklet provided by the researcher. In brief, diet encompasses a focus on minimally processed food, incorporating a wide variety of fruits, vegetables, legumes and wholegrains, whilst utilising olive oil as the main source of fat. They will be encouraged to eat more oily and white fish, with moderate consumption of nuts, poultry and dairy products, and low consumption of red/processed meat and alcohol.
  Participants in this group will also be performing home-based, equipment-free HIIT exercise for 20 minutes, 3 times a week for the duration of the 8-weeks, achieving ≥80% of predicted heart rate maximum (HRmax; 220-age) during the high-intensity intervals. Participants are also required to exercise at least 17 out of 20 on the Rate of Perceived Exertion (RPE) scale.
  Interventions: Other: Exercise and Mediterranean Diet (Ex + MedDiet)
- Control (No Intervention): Participants will be asked to maintain their diet and physical activity levels throughout the 8 weeks.

INTERVENTIONS:
Other: Exercise Only (Ex only) — Unsupervised, home-based, equipment-free high-intensity interval training of 20 minutes exercise performed 3 times a week, for a duration of 8-weeks. Participants will perform exercises to their own suitability in a progressive manner throughout the 8-weeks. Exercises will be exerted at least ≥80% of predicted heart rate maximum (HRmax; 220-age) during the high-intensity intervals, as well as at least 17 out of 20 Rate of Perceived Exertion on the Borg Scale.
  Arms: Exercise only (Ex only)
Other: Exercise and Mediterranean Diet (Ex + MedDiet) — Participants in Ex+MedDiet arm adhere to a non-caloric restrictive Mediterranean diet throughout the 8-weeks comprising of a diet encompassing a focus on minimally processed food, incorporating a wide variety of fruits, vegetables, legumes and wholegrains, whilst utilising olive oil as the main source of fat. They will be encouraged to eat more oily and white fish, with moderate consumption of nuts, poultry and dairy products, and low consumption of red/processed meat and alcohol.
  Participants will also perform unsupervised, home-based, equipment-free high-intensity interval training of 20 minutes exercise performed 3 times a week, for a duration of 8-weeks. Participants will perform exercises to their own suitability in a progressive manner throughout the 8-weeks. Exercises will be exerted at least ≥80% of predicted heart rate maximum (HRmax; 220-age) during the high-intensity intervals, as well as at least 17 out of 20 Rate of Perceived Exertion on the Borg Scale.
  Arms: Exercise and Mediterranean Diet (Ex + MedDiet)

SUMMARY:
This study proposes to examine the independent and combined effects of an 8-week home-based, equipment-free HIIT exercise intervention with/without Mediterranean diet through ghrelin-mediated alteration in overweight and obese metabolic women to improve cardiovascular-risk related markers and metabolic risk factors.

DETAILED DESCRIPTION:
This is a randomised-controlled study investigating the independent and combined effects of a home-based, equipment-free high intensity interval training (HIIT) exercise intervention with/without the Mediterranean diet (MedDiet) through ghrelin-mediated alteration on body composition, cardiovascular risk-related markers, metabolic markers and obesity-related hormones in postmenopausal women. The intervention will last for 8-weeks, with three arms comprising of 1) exercise only (Ex); 2) exercise and MedDiet (Ex+MedDiet); 3) control (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Participants >45-65 years of age
* Body mass index (BMI) >25.0 - 35.0
* Postmenopausal (with spontaneous amenorrhea for the last 12 months)
* Healthy (no known diseases)
* Physically inactive (IPAQ score - category I and not engaged in at least 60 min/week of structured exercise during the previous 6 months)
* Generally well enough to exercise.

Exclusion Criteria:

* Any inclusion criteria not met
* Abnormal ECG
* Current smokers
* Current or history of substance abuse and/or excess alcohol intake
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* On hormone therapy for <6 months
* Prescribed anti-hypertensive or beta-blocker medication

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Visceral adiposity index (VAI) | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). VAI calculated based on their waist circumference, BMI, triglycerides and HDL cholesterol levels. Waist circumference will be recorded in centimetres. BMI will be combined based on weight (kilograms) and height (metres) as kg/m^2. Triglycerides and HDL cholesterol levels will be assessed from fasting blood collected from the antecubital vein via venepuncture. Triglycerides and HDL will be recorded in mmol/L.
Inflammatory markers | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). IL-6, CRP, IL-10, TNF-α will be assessed from fasting blood collected from the antecubital vein via venepuncture.
Blood lipid levels | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). Triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol will be assessed from fasting blood collected from the antecubital vein via venepuncture. All blood lipids will be recorded in mmol/L.
Blood pressure | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). Systolic and diastolic blood pressure will be obtained from the participant's left arm after resting for at least 10 minutes. Blood pressure will be recorded in mmHg.
Insulin resistance index (HOMA-IR) | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). Calculated based on blood glucose levels (mmol/L) and insulin (pmol/L) from fasting blood collected from the antecubital vein via venepuncture.

SECONDARY OUTCOMES:
Circulatory levels of ghrelin | Baseline to 8 weeks
  Assessed at baseline and post-intervention (Week 1 and Week 8). Fasting circulatory levels of acyl and des-acyl ghrelin will be assessed from fasting blood collected from the antecubital vein via venepuncture. Acyl and des-acyl ghrelin will be recorded in pg/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided